CLINICAL TRIAL: NCT06139666
Title: The Effect of Liposomal Bupivacaine Nerve Block on Postoperative Pain After a Rotator Cuff Repair or Shoulder Arthroscopy
Brief Title: The Effect of Liposomal Bupivacaine Nerve Block (Exparel) in Rotator Cuff Surgery
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: The Cooper Health System (Other)
Responsible Party: Principal Investigator, Catherine Fedorka MD, Orthopaedic Surgeon, Assistant Professor of Orthopaedic Surgery, Assistant Program Director, Orthopaedic Surgery Residency Program, The Cooper Health System
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB 19-063
Record Dates: First submitted 2023-07-26; First posted 2023-11-18 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Rotator Cuff Tears; Postoperative Pain; Opioid Use
Keywords: Rotator Cuff Repair; Postoperative Pain Control; Orthopedic Surgery; Anesthesia; Nerve block; bupivacaine; Liposomal Bupivacaine
MeSH Terms: conditions — Rotator Cuff Injuries; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Prospective, double-blinded (surgeon and patient) randomized therapeutic trial
Who Masked: Participant, Investigator
Masking Description: Papers with equal numbers of either "E" for Exparel or "B" for Bupivacaine will be allocated to envelopes and shuffled for randomization. At the time of selection, the patient will be identified and allocated to their respective group dependent on what letter they get. This will take place in the preoperative visit and will be communicated to the anesthesia team prior to block taking place by the data spreadsheet so that the surgeon will be blinded to what treatment took place.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control- Bupivacaine Alone (Active Comparator): patients will receive a standard interscalene block with bupivacaine alone (25 cc of bupivacaine)
  Interventions: Drug: Bupivacaine Injectable Solution
- Study- Exparel (Experimental): patients will receive an interscalene block with Exparel solution, which is an extended-release formulation of bupivacaine consisting of 10cc liposomal bupivacaine mixed with 15cc bupivacaine. This is approved and used at the study institution
  Interventions: Drug: Exparel Injectable Solution

INTERVENTIONS:
Drug: Exparel Injectable Solution — Patients randomized to this arm will receive an interscalene block with Exparel solution, an extended-release formulation of bupivacaine (10cc liposomal bupivacaine + 15cc bupivacaine), approved for use at the study institution. This will be administered preoperatively on the day of surgery. The anesthesiologist administering the injection will be not be blinded to the mixture of injections (the surgeon and the patient will), which will be designated and randomized prior to administration. They will order and draw up the medication as they have been previously with no change in the standard of care.
  After surgery, the patient will be asked to keep a daily log of their pain scores, and the amount of narcotics will be counted by the physician at the first postoperative visit. The block would have been offered to the patient even if they are not part of the study. No additional visits are required. The only difference is the journal with pain score surveys and the pill count.
  Arms: Study- Exparel
Drug: Bupivacaine Injectable Solution — Patients randomized to this arm will receive a standard interscalene block consisting of 25 cc of bupivacaine alone. This will be administered preoperatively on the day of surgery.
  The anesthesiologist administering the injection will not be blinded to the mixture of injections (the surgeon and the patient will), which will be designated and randomized prior to administration. They will order and draw up the medication as they have been previously with no change in the standard of care.
  After surgery, the patient will be asked to keep a daily log of their pain scores, and the amount of narcotics will be counted by the physician at the first postoperative visit. The block would have been offered to the patient even if they are not part of the study. No additional visits are required. The only difference is the journal with pain score surveys and the pill count.
  Arms: Control- Bupivacaine Alone

SUMMARY:
The goal of this clinical trial is to investigate if there is a difference in pain after an arthroscopic rotator cuff surgery when a nerve block is performed with liposomal bupivacaine versus the standard treatment of bupivacaine alone.

The main question aims to answer if patients who receive liposomal bupivacaine have better pain control and lower postoperative opioid consumption compared to bupivacaine alone.

Participants be randomized to either the control group to receive a standard interscalene block with bupivacaine (25 cc of bupivacaine) or the experimental group to receive similar dosing of liposomal bupivacaine mixed with bupivacaine (10cc liposomal bupivacaine + 15cc bupivacaine). Data will be prospectively collected and the data from the experimental group will be compared to the control group at the completion of the study period.

DETAILED DESCRIPTION:
Nerve blocks are typically performed for shoulder surgery for perioperative pain control. This is performed in the shoulder using an interscalene block, which is localized between the anterior and middle scalene muscles in the neck and provides analgesia to the clavicle, shoulder and its capsule and some to the arm. Using this method allows for conscious sedation to be used over general anesthesia, mitigating the dangers associated with the latter, and also comes with the added benefit of providing improved postoperative analgesia.

Bupivacaine is the medication that is typically used for these procedures to provide the analgesia in these sensory patterns. It works by binding to the intracellular portion of voltage-gated sodium channels, preventing depolarization of the nerve and subsequently inhibiting transmission of nerve signals. Typical interscalene blocks have been shown to have pain control for 6-8 hours and have an effect decreasing opioid usage for up to 24 hours. Liposomal bupivacaine, trade name Exparel, was recently introduced as an alternative to drugs such as bupivacaine, but boasting a longer duration of action. In Exparel, bupivacaine is stored in liposomes, which allows for a controlled and longer duration of release of the analgesia-producing molecules. This allows nerve blockades to last longer, allowing for longer prevention of neurotransmitter release. It was initially only approved for local infiltration, most notably in the joint capsule for a total knee arthroplasty. Recently however, it was FDA approved for interscalene blocks, opening up a new avenue for pain control modalities. No studies have yet been performed comparing the difference in analgesia provided by liposomal bupivacaine compared to bupivacaine alone in the context of interscalene blocks in rotator cuff surgery

Nerve blocks with local anesthetics has been proven safe and effective for perioperative pain control. With recent talks of healthcare providers decreasing narcotic usage postoperatively in an effort to prevent opiate addiction, longer acting nerve blocks are becoming more and more appealing. By increasing the duration of a nerve blockade, postoperative narcotic use may be significantly decreased, with minimal risk of harm to the patient.

This is a prospective, double-blinded (surgeon and patient) randomized therapeutic trial. Patients will either receive a standard interscalene block with bupivacaine (25 cc of bupivacaine) or will receive similar dosing of liposomal bupivacaine mixed with bupivacaine (10cc liposomal bupivacaine + 15cc bupivacaine), which has recently been approved and instituted. These blocks (both) are currently in practice at the study institution and the decision of which to use is currently up to the anesthesiologist. It is current practice that every patient undergoing a rotator cuff surgery is offered a nerve block. Data will be prospectively collected and the data from the experimental group will be compared to the control group at the completion of the study period.

Patents will present for surgery and follow up postoperatively as they would routinely for rotator cuff surgery or shoulder arthroscopy. The anesthesiologist administering the injection will be not be blinded to the mixture of injection (the surgeon and the patient will), which will be designated and randomized prior to administration. They will order and draw up the medication as they have been previously with no change in the standard of care.

When discharged home, patients will be asked to keep a log of their narcotic consumption, as well as bringing in their prescription vial to the postoperative follow up and also logging other medications that are consumed during this time period. They will also be asked to log their pain scores in the form of a standardized VAS pain scale form that they will fill out daily until their first follow up visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients above 18 years of age
* Undergoing rotator cuff surgery or shoulder arthroscopy using an interscalene block

Exclusion Criteria:

* Patients with preexisting chronic obstructive pulmonary disease (COPD) or respiratory issues precluding the use of an interscalene block
* Pregnant women, women nursing infants
* Patients with preexisting liver disease
* Patients unwilling to have interscalene block performed
* Patients allergic to bupivacaine, liposomal bupivacaine, or any ingredients contained within the two drugs listed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2019-07-11 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Use of pain medications | 2 week postoperative visit
  Patients will be asked to bring their bottle of pain medication prescribed after surgery to their first office visit so a narcotic pill count can be performed. Patients will record their pain pill consumption every day for 2 weeks in a study journal. The journal containing the pill count will be collected at the 2 week visit in the office. Opioid consumption will be quantified as milligram of opioid equivalents (MME).

SECONDARY OUTCOMES:
Pain severity | Every day for the first 2 weeks, and a one-time survey at the 6 week and 12 week visit.
  Patients will rate their pain using the VAS pain scale survey. The visual analog scale (VAS) is a pain rating scale first used by Hayes and Patterson in 1921. Scores are based on self-reported measures of symptoms that are recorded with a single handwritten mark placed at one point along the length of a 10-cm line that represents a continuum between the two ends of the scale-"no pain" on the left end (0 cm) of the scale and the "worst pain" on the right end of the scale (10 cm). These results will be recorded every day for the first 2 weeks in a study journal. The journal containing the VAS scores will be collected at the 2 week visit in the office. The VAS will be administered again at the 6 week and 12 week visit.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine J Fedorka, MD, Principal Investigator — The Cooper Health System
Locations (1):
- Cooper University Hospital, Camden, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim DH, Liu J, Beathe JC, Lin Y, Wetmore DS, Kim SJ, Haskins SC, Garvin S, Oxendine JA, Ho MC, Allen AA, Popovic M, Gbaje E, Wu CL, Memtsoudis SG. Interscalene Brachial Plexus Block with Liposomal Bupivacaine versus Standard Bupivacaine with Perineural Dexamethasone: A Noninferiority Trial. Anesthesiology. 2022 Mar 1;136(3):434-447. doi: 10.1097/ALN.0000000000004111. PMID 35041742
- [Background] Wiederhold BD, Garmon EH, Peterson E, Stevens JB, O'Rourke MC. Nerve Block Anesthesia. 2023 Apr 29. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK431109/ PMID 28613761
- [Background] Lonner JH, Scuderi GR, Lieberman JR. Potential utility of liposome bupivacaine in orthopedic surgery. Am J Orthop (Belle Mead NJ). 2015 Mar;44(3):111-7. PMID 25750943
- [Background] Vyas KS, Rajendran S, Morrison SD, Shakir A, Mardini S, Lemaine V, Nahabedian MY, Baker SB, Rinker BD, Vasconez HC. Systematic Review of Liposomal Bupivacaine (Exparel) for Postoperative Analgesia. Plast Reconstr Surg. 2016 Oct;138(4):748e-756e. doi: 10.1097/PRS.0000000000002547. PMID 27673545
- [Background] Kaye AD, Armstead-Williams C, Hyatali F, Cox KS, Kaye RJ, Eng LK, Farooq Anwar MA, Patel PV, Patil S, Cornett EM. Exparel for Postoperative Pain Management: a Comprehensive Review. Curr Pain Headache Rep. 2020 Oct 23;24(11):73. doi: 10.1007/s11916-020-00905-4. PMID 33098008
- [Derived] Fedorka CJ, Tornberg HN, Rivera-Pintado C, Gentile PM, Russo D, Boniello M, Hunter K, Desai R, Soni D, Kleiner MT, Dodson G. Liposomal Bupivacaine + Bupivacaine Versus Bupivacaine Interscalene Nerve Block Effect on Pain After Rotator Cuff Repair: A Randomized Control Trial. J Am Acad Orthop Surg. 2025 Dec 24. doi: 10.5435/JAAOS-D-25-01002. Online ahead of print. PMID 41468585